CLINICAL TRIAL: NCT05914454
Title: Efficacy and Safety of Anakinra in Acute Respiratory Distress Syndrome
Acronym: ESKA
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Azienda Sanitaria-Universitaria Integrata di Udine (Other)
Collaborators: University of Udine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 4381
Record Dates: First submitted 2023-06-13; First posted 2023-06-22 (Actual); Last update posted 2023-06-22 (Actual); Status verified 2023-06

CONDITIONS: Acute Respiratory Distress Syndrome
Keywords: IL-1; anakinra; acute respiratory distress syndrome; lung
MeSH Terms: conditions — Respiratory Distress Syndrome | interventions — Interleukin 1 Receptor Antagonist Protein

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- anakinra (Experimental): anakinra 100 mg/day for 14 consecutive days
  Interventions: Drug: Anakinra 100Mg/0.67Ml Inj Syringe
- standard of care (No Intervention)

INTERVENTIONS:
Drug: Anakinra 100Mg/0.67Ml Inj Syringe — anakinra 100 mg per day for 14 days
  Arms: anakinra

SUMMARY:
Acute Respiratory Distress Syndrome (ARDS) is a life-threatening condition characterized by acute respiratory failure with hypoxemia, noncardiogenic or non-fluid overload pulmonary edema, bilateral diffuse opacities on chest radiograph in the presence of a predisposing factor.

In ARDS there is activation of the inflammatory cascade which is very intense and persistent in the severe types. It was highlighted that the inflammatory cytokines in patients with ARDS or sepsis is similar to that observed in COVID-19 positive patients.

Emerging therapies include immunomodulation and the administration of mesenchymal stem cells for the modulation of lung repair through the release of cytokines and growth factors that modulate the local inflammatory response.

Regardless of the cause of ARDS, the severity of the inflammatory state and fibroproliferative evolution have been shown to be independent predictors of survival and ventilator dependence. Patients suffering from severe forms of ARDS in fact require prolonged mechanical ventilation, which exposes them to ventilator-associated pneumonia (VAP) and the onset of multiorgan insufficiency. The hyperinflammatory state underlying ARDS predisposes to pulmonary fibroproliferation, which in turn increases susceptibility to ventilator dependence and increases the risk of MOF and death. For this reason, the rationale in the use of anakinra is to limit the inflammatory process of ARDS as early as possible, avoiding the progression of lung damage.

ELIGIBILITY:
Inclusion Criteria:

* Patients admitted to intensive care unit diagnosed within 48 hours of moderate-severe ARDS (PaO2/FiO2 < 200, PEEP ≥ 5 cmH2O) and requiring intubation and mechanical ventilation;
* Berlin clinical criteria for definition of ARDS: onset within 1 week of initial lesion or new or worsening respiratory symptoms, bilateral opacities not fully explained by effusions, lobar or lung collapse or nodules, respiratory failure not fully explained by heart failure or fluid overload
* ARDS-like clinical-laboratory profile, defined by at least one of the following criteria:

  * high plasma levels of inflammatory biomarkers (e.g. IL-6 > 80 pg/ml, CRP > 250 mg/l)
  * dependence on vasopressors (of any type and at any dosage for at least one hour of treatment)
  * reduction of bicarbonatemia (< 18 mMol/L) or hyperlactacidemia (> 4 mMol/L)
* Informed consent for participation in the study
* Negative swab for COVID-19.

Exclusion Criteria:

* Pregnant or lactating patients;
* Hypersensitivity to the active substance or to any of the excipients or to proteins derived from Escherichia Coli;
* Concomitant treatment with anti-TNF-alpha or other biotechnological agent;
* Neutropenia (neutrophils < 1.5 x 109/L);
* Pre-existing malignancies;
* Moderate to severe renal insufficiency, creatinine clearance < 60 ml/minute.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2023-05-19 (Actual); Primary Completion 2025-06-19 (Estimated); Study Completion 2025-09-19 (Estimated)

PRIMARY OUTCOMES:
Assessment of ventilation-free days | 28 days
  The calculation will take place from the day of extubation to the 28th day of hospitalization. Patients who die before ventilator weaning will be considered as having 0 days off ventilation. The calculation of the days free from ventilation will be calculated as follows: 28 - number of days of ventilation.

CONTACTS AND LOCATIONS:
Overall Officials: Tiziana Bove, MD, PhD, Principal Investigator — Azienda Sanitaria Universitaria Friuli Centrale
Locations (1):
- Azienda Sanitaria Universitaria, Udine, Italy

IPD SHARING:
Plan to Share IPD: No